CLINICAL TRIAL: NCT03159429
Title: Nasal Ventilation Versus Voluntary Hypoventilation in the Rehabilitation of Hyperventilation Syndrome: a Randomized, Controlled Trial
Brief Title: Nasal Ventilation Versus Voluntary Hypoventilation in the Rehabilitation of Hyperventilation Syndrome
Acronym: RehabSHV
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Staff no longer available.
Sponsor: University Hospital, Montpellier (Other)
Collaborators: APARD Fonds de dotation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9796; 2017-A00554-49 (Other: RCB number)
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Hyperventilation Syndrome
Keywords: Dyspnea; Rehabilitation of olfaction; Hyperventilation syndrome
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Intervention Model Description: The included population will be randomized into two parallel groups. One group will be assigned the experimental intervention. The other group will be assigned standard care. Outcomes will be compared between the two randomized groups.
Masking Description: Given that the experimental and comparator interventions concern behaviour and exercises, it is not possible to blind participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): Patients randomized to this arm will participate in the new rehabilitation programme.
  Intervention: Nasal breathing rehabilitation
  Interventions: Behavioral: Nasal breathing rehabilitation
- Comparator arm (Active Comparator): Patients randomized to this arm will participate in the usual rehabilitation programme.
  Intervention: Standard rehabilitation
  Interventions: Behavioral: Standard rehabilitation

INTERVENTIONS:
Behavioral: Standard rehabilitation — The patient will participate in a therapeutic education programme consisting of 4 visits (days 1 +- 14, 21 +- 14, 61 +- 14 and 90 +-14) representing usual procedures, which include: maintaining a diary, breathing coordination excercises, voluntary control of breathing rate, releasing contracted muscles, posture harmonization, a six minute walking test, and walking up four flights of stairs.
  Arms: Comparator arm
Behavioral: Nasal breathing rehabilitation — The patient will participate in a therapeutic education programme consisting of 4 visits (days 1 +- 14, 21 +- 14, 61 +- 14 and 90 +-14) representing the experimental procedures, which include: maintaining a diary, evaluating nasal breathing by the nostril-alternating technique according to Anuloma Viloma Pranayama Yoga, releasing contracted muscles, posture harmonization, a six minute walking test, and walking up four flights of stairs.
  Arms: Experimental arm

SUMMARY:
The main objective of this study is to measure the effect (at 3 months) of dyspnea control rehabilitation with nasal ventilation versus standard rehabilitation, in dyspneic patients with hyperventilation syndrome.

DETAILED DESCRIPTION:
Hyperventilation syndrome (SHV) is a complex disorder of adaptation of ventilation to exercise. This is a frequent reason for consultation because it is associated with major symptoms, which can be a source of sometimes heavy exploration and wandering. The breathless patient reduces his activity and enters the vicious circle of deconditioning. The principal clinical symptom in this pathology is the dyspnea with hypocapnia. The diagnosis is based on quality of life questionnaires and provocation tests, such as stress testing. When hypocapnia becomes chronic, a disturbance of breathing control sets in.

In SHV therapy, control of ventilation to exercise is recommended in the first line. It aims to slow the respiratory rate or tidal volume with, for example, techniques of voluntary hypoventilation and abdominal ventilation. But the evidence of literature is lacking to recommend a particular technique. Given the implication of the dysfunction of the nose, of non-unicist and often multifactorial origin in the respiratory pathologies, one of the possibilities of intervention is to reeducate the patient to the nasal ventilation.

Our rehabilitation of nasal ventilation is based on the clinical observation of hyperventilation dyspnea. During breathlessness breathing is essentially oral. It is a natural mechanism of adaptation that responds to the metabolic demand, which is far too present in the hyperventilation syndrome. From our therapeutic experience, the hypothesis is that the work on nasal ventilation can provide the necessary elements for the correction of SHV. The importance of the nasal breath in managing emotions and effort in sport is already considered.

This study will evaluate pathophysiological and clinical parameters effets of rehabilitation of nasal ventilation compared to those of the technique of voluntary hypoventilation (ThV) which is the conventional management of patients with SHV.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his / her free and informed consent and signed the consent
* The patient must be a member or beneficiary of a health insurance program
* The patient is available for 3 months of follow-up
* The patient has at least two of the following clinical symptoms consistent with hyperventilation sydrome: dyspnea, chest pain or pressure, visual blurring, dizziness, a sensation of abdominal swelling, tingling in the fingers, stiffness in the fingers or arms, tingling sensation around the mouth, cold or moist hands, tension or anxiety
* Resting hypocapnia defined by a PaCO2 <38 mmHg and a normal O2 alveolo-arterial gradient D (A-a) O2
* Absence of significant obstructive or restrictive pathology according to respiratory function tests
* Absence of indirect signs of pulmonary arterial hypertension according to echocardiography
* Absence of alteration of gas exchange on maximum cardiopulmonary stress test (elevation of gradient D (A-a) O2 > 35 mmHg at peak stress)
* At least 2 of the following criteria: (i) a Nijmegen questionnaire score > 23, (ii) the recurrence of at least two common symptoms during the maximum cardiopulmonary stress test, (iii) delayed return of PETCO2 (partial pressure of end-tidal carbon dioxide) to its basal value (> 5 minutes)

Exclusion Criteria:

* The subject is participating in another study
* The subject is in an exclusion period determined by a previous study
* The subject is under judicial protection, or is an adult under any kind of guardianship
* The subject refuses to sign the consent
* It is impossible to correctly inform the subject
* The subject cannot fluently read French
* The patient is pregnant
* The patient is breastfeeding
* The subject has a contra-indication (or an incompatible drug association) for a treatment required during this study (a priori, there are no contra-indicated drugs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Change in Dyspnea at VO2max | Change between Day 0 and Day 90 +- 30
  Dyspnea measured at the first VO2max during a maximal cardio-pulmonary effort test. Dyspnea is measured using a visual analog scale.

SECONDARY OUTCOMES:
Time to start of mouth-breathing during exercise test | Change between Day 0 and Day 90 +- 30
  The delay of onset of oral ventilation during walking and / or on ergocycle
The SNOT22 questionnaire score | Change between Day 0 and Day 90 +- 30
  The SNOT22 questionnaire score
Ventilation during isowork | Change between Day 0 and Day 90 +- 30
  (Ventilation equivalents V'E / V'O2 and V'E / V'CO2)
PACO2 at rest | Change between Day 0 and Day 90 +- 30
  PAC02 = Partial pressure of carbon dioxide in arterial blood
pH at rest | Change between Day 0 and Day 90 +- 30
  pH at rest
PaO2 at rest | Change between Day 0 and Day 90 +- 30
  PaO2 = Partial pressure of oxygen in arterial blood
PACO2 at maximum effort | Change between Day 0 and Day 90 +- 30
  PAC02 = Partial pressure of carbon dioxide in arterial blood
pH at maximum effort | Change between Day 0 and Day 90 +- 30
  pH at maximum effort
PaO2 at maximum effort | Change between Day 0 and Day 90 +- 30
  PaO2 = Partial pressure of oxygen in arterial blood
Breathing rates during excerise testing | Change between Day 0 and Day 90 +- 30
  breaths per minute
Transcutaneous oximetry | Change between Day 0 and Day 90 +- 30
  tcpO2
Distance walked during 6 minute walking test | Change between Day 0 and Day 90 +- 30
  Distance walked during 6 minute walking test
Maximum rate of oxygen consumption | Change between Day 0 and Day 90 +- 30
  VO2max
Maximum dyspnea values | Change between Day 0 and Day 90 +- 30
  Dyspnea is measured using visual analogue scales
Dyspnea threshold during exercise testing | Change between Day 0 and Day 90 +- 30
  Dyspnea is measured using visual analogue scales
The slope of the equation VE=f(PETCO2) | Change between Day 0 and Day 90 +- 30
  VE = expiratory ventilation ; PETCO2 = end tidal carbon dioxide tension
PETCO2 value when VE = 0 | Change between Day 0 and Day 90 +- 30
  VE = expiratory ventilation ; PETCO2 = end tidal carbon dioxide tension
the equation P0.1=f(PETCO2) | Change between Day 0 and Day 90 +- 30
  P0.1 = occlusion pressure; PETCO2 = end tidal carbon dioxide tension
Dyspnea measured using the MRC scale | Change between Day 0 and Day 90 +- 30
  Dyspnea measured using the Medical Research Council scale
Nijmegen questionnaire score | Change between Day 0 and Day 90 +- 30
  Nijmegen questionnaire score
SF36 questionnaire score | Change between Day 0 and Day 90 +- 30
  SF36 questionnaire score
VQ-11 questionnaire score | Change between Day 0 and Day 90 +- 30
  VQ-11 questionnaire score
HAD questionnaire score | Change between Day 0 and Day 90 +- 30
  HAD questionnaire score

CONTACTS AND LOCATIONS:
Overall Officials: Florence Pourias Laborde, DE, Study Director — University Hospital, Montpellier
Locations (1):
- Montpellier University Hospital, Montpellier, France